CLINICAL TRIAL: NCT04110860
Title: Clinical Evaluation of a Formulated Nanoemulsion for Topical Application
Brief Title: Clinical Assessment of Voriconazole Self Nano Emulsifying Drug Delivery System Intermediate Gel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sara Botros (Other)
Responsible Party: Sponsor-Investigator, Sara Botros, demonstrator, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCZSaraSNEDDS
Record Dates: First submitted 2019-09-28; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Tinea Versicolor
MeSH Terms: conditions — Tinea Versicolor

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- once daily application (Experimental): the gel is applied to the affected areas once daily for one week followed by a follow-up visit to reassess the case. if complete cure is achieved, stop application. if not, repeat for one more week and then reassess.
  Interventions: Drug: voriconazole gel once daily
- twice daily application (Experimental): the gel is applied to the affected areas twice daily for one week followed by a follow-up visit to reassess the case. if complete cure is achieved, stop application. if not, repeat for one more week and then reassess.
  Interventions: Drug: voriconazole gel twice daily
- placebo (Placebo Comparator): the gel is applied to the affected areas twice daily for one week followed by a follow-up visit to reassess the case. if complete cure is achieved, stop application. if not, repeat for one more week and then reassess.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: voriconazole gel once daily — voriconazole is incorporated into a nanoemulsion intermediate gel state then applied on the affected areas once daily
  Arms: once daily application
Drug: voriconazole gel twice daily — voriconazole is incorporated into a nanoemulsion intermediate gel state then applied on the affected areas twice daily
  Arms: twice daily application
Drug: placebo — the same procedure as before is used to prepare the nanoemulsion intermediate gel but the active ingredient, voriconazole, is not added then applied twice daily in the same manner
  Arms: placebo

SUMMARY:
Clinical study for the developed voriconazole self nano emulsifying drug delivery system intermediate gel was conducted on 30 patients with tinea versicolor infection.

DETAILED DESCRIPTION:
The clinical work has been carried out in accordance with The Code of Ethics of the World Medical Association for experiments involving humans. The study was conducted on 30 patients (10 to 60 years old) with tinea versicolor attending the dermatology department outpatient clinic of Minia University Hospital. Local institutional review board approval was obtained for this study (ethical approval number is 24/18). Pregnant or lactating females and Immunocompromized patients. The patients were then divided into 3 groups, placebo group, group A and group B, consisting of 10 patients each. The placebo group received unmedicated formulation, Group A received the medicated formulation once daily and group B were treated twice daily. An informed consent has been obtained from all patients enrolled in the study for photography and treatment. History and general local examination were performed for all patients.The patients were clinically examined under normal light and using wood's lamp and cello-tape test was performed to confirm infection after determining the type of infection and in some cases scrapes were taken to detect infection in clinically indefinite cases and stained using potassium hydroxide 20% then examined for presence of fungal elements. Treatment was performed by applying the gel once or twice daily until full recovery was achieved with follow up once a week to reassess the condition. The clinical improvement of the patients, patient satisfaction and length of treatment were assessed. It was rated by both patient and physician as excellent, good, fair or poor according to the following criteria. Excellent: both the patient and the physician agreed that the result was satisfactory. Good: the result although acceptable was not quite up to expectations, but the physicians were pleased with the outcome. Fair: the improvement was evaluated by both the patient and the physician to be less than expected but still with some improvement. Poor: unsatisfactory results to the patient and /or the physician. All adverse effects were checked during study.High resolution digital photographs were taken for lesions of all patients using identical camera folder setting before starting treatment, on each follow up visit and after complete recovery. Clinical improvement was evaluated by physicians. The criteria for evaluations using a quartile grading scale were: 0=no improvement. 1=mild (percent improvement, less than 25%), 2=moderate (percent improvement 25-49%), 3=good (percent improvement 50-74%), 4=excellent (percent improvement equal to or more than 75%). In addition, a patient satisfaction score was rated using the following scale, A. satisfied, B.

ELIGIBILITY:
Inclusion Criteria:

* Tinea Versicolor infection

Exclusion Criteria:

* concomitant treatment with other medications for the same condition being studied, TVC.
* pregnancy
* lactation
* immunocompromised patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
complete cure | 1-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sara R Botros, bachelor of clinical pharmacy, Principal Investigator — Minia University
Locations (1):
- Minia University hospital, Minya, Minya Governorate, Egypt